CLINICAL TRIAL: NCT07358559
Title: Teaming Researchers Up With Stakeholders to Test Trustworthy Engagement and Measures
Brief Title: Scale Development for Organizational Trustworthiness
Acronym: TRUST TEAM
Status: Not yet recruiting | Type: Observational
Sponsor: The Hastings Center for Bioethics (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY25090191
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Psychometric
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — This is not an intervention study.

SUMMARY:
The Teaming Researchers Up with Stakeholders to Test Trustworthy Engagement and Measure (TRUST TEAM) project seeks to better understand the role of organizational trustworthiness in the context of community-engaged research. At its core, how does organizational trustworthiness shape patients and other key stakeholders' involvement in community-academic research collaborations? What characteristics make an organization trustworthy and how does that strengthen relationships between academic organizations and community collaborators?

This project is creating a first-of-its-kind psychometrically sound measure of organizational trustworthiness.

ELIGIBILITY:
Inclusion Criteria:

* Community/Advocacy Leaders, Clinician Non-Researchers, Patient Stakeholders

Exclusion Criteria:

* Clinical Researchers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have been engaged as co-collaborates in community engaged research projects.
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Development of Organizational Trustworthiness Measure | April 2025 to October 2026
  Develop and test a measure of organizational trustworthiness

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Brown, PhD, MA, Principal Investigator — The Hastings Center for Bioethics

IPD SHARING:
Plan to Share IPD: No